CLINICAL TRIAL: NCT03562247
Title: Telenursing With or Without Remote Monitoring Compared to Usual Care for Patients Newly Diagnosed With Idiopathic Pulmonary Fibrosis.
Brief Title: Telenursing and Remote Monitoring in Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution and the study was closed with the IRB
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Lancaster, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tenure-1
Record Dates: First submitted 2018-06-14; First posted 2018-06-19 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Telenursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care of IPF (Active Comparator): Newly diagnosed patients will continue to receive excellent healthcare as currently given in management of the lung disease
  Interventions: Other: Usual Care of IPF
- Telenursing (Experimental): Patients will receive usual care with structured phone calls from the nurse practitioner and/or case manager occuring more frequently earlier in the diagnosis to help the patient and care giver understand all aspects of the disease and it time will evolve to managing symptoms outside of out-patient clinic visits.
  Interventions: Other: Usual Care of IPF; Other: Telenursing
- Telenursing and Remote Monitoring (Experimental): Patients will receive usual care with telenursing and will be given a hand held spirometer and puse oximeter and be asked to take daily measurements and report these via an electronic HIPAA approved secured platform for evaluation by the telenursing team.
  Interventions: Other: Usual Care of IPF; Other: Telenursing; Other: Telenursing and Remote Monitoring

INTERVENTIONS:
Other: Usual Care of IPF — standard of care given to patients with IPF
Other: Telenursing — scheduled phone calls with the patient and care giver
  Arms: Telenursing; Telenursing and Remote Monitoring
Other: Telenursing and Remote Monitoring — scheduled phone calls and home monitoring of physiologic parameters
  Arms: Telenursing and Remote Monitoring

SUMMARY:
Numerous studies show that remote monitoring and/or telenursing improves outcomes for patients especially those with chronic diseases. It is proposed that structured telenursing with non-invasive home monitoring of forced vital capacity and oxygen saturation in newly diagnosed patients with IPF will decrease hospitalizations for respiratory illness, increase compliance with therapies, and ultimately increase quality of life.

DETAILED DESCRIPTION:
Patients undergoing evaluation for and who are diagnosed with Idiopathic Pulmonary Fibrosis at Vanderbilt Medical Center from August 1, 2018, will be asked to participate. If agrees, and after signing the consent form, patients will be randomized into one of three arms: Usual Care, Usual Care with Telenursing, or Usual Care with Telenursing and Remote Monitoring. Patients will be asked to remain in the study for a minimum of three years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be newly diagnosed with IPF by a Vanderbilt pulmonologist according to the 2011 American Thoracic Society Guidelines. If the patient has been diagnosed by local pulmonologist and started on FDA-approved treatment, then must have been started on treatment within 6 months of Vanderbilt University Medical Center-based diagnosis.
2. Willingness to complete Quality of Life and Compliance Questionnaires at 6-month intervals either via an on-line process (RED Cap survey) or paper-based.
3. Willingness to participate in phone calls/video calls with the nurse practitioner or nurse case manager, if assigned to Arm 2 or Arm 3.
4. Willingness to complete and monitor daily health assessments, if assigned to Arm 3.
5. Willingness to share objective data via a provided electronic web-based portal, electronically via email, fax, or regular mail.
6. Willingness to notify, or allow notification, of study involvement with local pulmonary practices.

Exclusion Criteria:

1. Diagnosed with any other interstitial lung disease.
2. Diagnosed and began treatment > 6 months before the VUMC-based diagnosis date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Lancaster, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care of Idiopathic Pulmonary Fibrosis (IPF): Newly diagnosed patients will continue to receive standard of care in management of Idiopathic Pulmonary Fibrosis (IPF)
  Usual Care of IPF: Standard of care given to patients with IPF
- Telenursing: Patients will receive usual care with structured phone calls from the nurse practitioner and/or case manager occurring more frequently earlier in the diagnosis to help the patient and care giver understand all aspects of the disease and it time will evolve to managing symptoms outside of out-patient clinic visits.
  Usual Care of IPF: Standard of care given to patients with IPF
  Telenursing: Scheduled phone calls with the patient and care giver
Period: Overall Study
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Started | 10 | 11 | 10
Completed | 7 | 10 | 9
Not Completed | 3 | 1 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring | Total
Number analyzed (Participants) | 10 | 11 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants] — Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data not collected includes: Usual Care: Missing data from 4 participants / Telenursing: Missing data from 4 participants / Telenursing and Remote Monitoring: Missing data from 2 participants. Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
  Participants
    number analyzed (Participants) | 6 | 7 | 8 | 21
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 3 | 1 | 3 | 7
    >=65 years | 3 | 6 | 5 | 14
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data not collected includes: Usual Care: Missing data from 3 participants / Telenursing: Missing data from 4 participants / Telenursing and Remote Monitoring: Missing data from 2 participants. Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
  Participants
    number analyzed (Participants) | 7 | 7 | 8 | 22
    Female | 3 | 3 | 3 | 9
    Male | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data not collected includes: Usual Care: Missing data from 3 participants / Telenursing: Missing data from 1 participant / Telenursing and Remote Monitoring: Missing data from 1 participant. Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
  Participants
    number analyzed (Participants) | 7 | 10 | 9 | 26
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 7 | 7 | 8 | 22
    Unknown or Not Reported | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data not collected includes: Usual Care: Missing data from 3 participants / Telenursing: Missing data from 1 participant / Telenursing and Remote Monitoring: Missing data from 1 participant. Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
  Participants
    number analyzed (Participants) | 7 | 10 | 9 | 26
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 0 | 1
    White | 7 | 6 | 8 | 21
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: The Number Hospitalization Events Resulting From a Respiratory Illness
Description: The number hospitalization events resulting from a respiratory illness
Time Frame: Baseline to 21 months
Measure: Number; unit: Events
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 10 | 9
Events | 1 | 0 | 0

2. Secondary Outcome: The Number of Respiratory Events That Indicate a Worsening of Idiopathic Pulmonary Fibrosis (IPF)
Description: The number of respiratory events that indicate a worsening of Idiopathic Pulmonary Fibrosis (IPF)
Time Frame: Baseline to 21 months
Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data was not collected for 3 participants in the Telenursing arm: Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
Measure: Number; unit: Events
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 7 | 9
Events
  5% decline in home FVC | 0 | 0 | 0
  4 percentage points decline in home saturation | 0 | 0 | 0
  respiratory infection | 0 | 0 | 1
  pneumonia | 0 | 0 | 0
  pneumothorax | 0 | 0 | 0
  pleural effusion | 0 | 0 | 0
  pulmonary embolus | 1 | 0 | 0
  >= 5% decline in clinic FVC (from last visit) | 3 | 0 | 1
  >= 10% decline in clinic FVC (from last visit) | 2 | 0 | 1
  >= 5% decline in clinic FVC (from one year ago) | 1 | 0 | 0
  >= 10% decline in clinic FVC (from one year ago) | 4 | 1 | 0

3. Secondary Outcome: The Number of Acute Exacerbations of Idiopathic Pulmonary Fibrosis (IPF)
Description: The Number of Acute Exacerbations of IPF
Time Frame: Baseline to 21 months
Measure: Number; unit: number of events
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 10 | 9
number of events | 0 | 0 | 0

4. Secondary Outcome: The Number of Days From Idiopathic Pulmonary Fibrosis (IPF) Diagnosis to First Hospitalization for Respiratory Illness
Description: The total combined number of days for all participants in each arm from the date of IPF diagnosis to the date of first hospitalization for respiratory illness.
Time Frame: Baseline to 21 months
Measure: Number; unit: days
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 10 | 9
days | 367 | NA — There were no hospitalization events for respiratory illness reported in the Telenursing Arm. As a result, data entry for this field is NA (not applicable). | NA — There were no hospitalization events for respiratory illness reported in the Telenursing and Remote Monitoring Arm. As a result, data entry for this field is NA (not applicable).

5. Secondary Outcome: The Severity of Dyspnea as Measured by the Modified Medical Research Council (mMRC) Dyspnea Scale
Description: Dyspnea (shortness of breath) was assessed using the mMRC, a single item (0-4) scale assessing current level of dyspnea. The mMRC comprised of five statements that describe almost the entire range of respiratory disability from none (Grade 0) to almost complete incapacity (Grade 4). The mMRC categorized participants into low dyspnea (Grades 0-1) and high dyspnea (Grades 2-4).
Time Frame: Baseline to 21 months
Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data was not collected for this outcome measure for 1 participant in the Telenursing and Remote Monitoring arm. Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 10 | 8
score on a scale
  Baseline: number analyzed (Participants) | 7 | 6 | 0
  Baseline | 1.5 (0.57) | 1 (1.09) |
  Visit 2 (3 months): number analyzed (Participants) | 2 | 3 | 4
  Visit 2 (3 months) | 1.5 (0.70) | 0.66 (0.57) | 1.5 (1.29)
  Visit 3 (9 months): number analyzed (Participants) | 2 | 1 | 3
  Visit 3 (9 months) | 3 (1.41) | 2 (0) | 0.33 (0.57)
  Visit 4 (15 months): number analyzed (Participants) | 0 | 0 | 0
  Visit 5 (21 months): number analyzed (Participants) | 0 | 0 | 1
  Visit 5 (21 months) |  |  | 0 (0)

6. Secondary Outcome: The Severity of Depression as Measured by the Adapted Mental Health America Depression Screening Tool
Description: The adapted Mental Health America Depression Screening Tool is an 8 question self-administered questionnaire that scores patient-reported symptoms of depression. The possible score for each question ranges from 0-3. The total questionnaire score range is 0-24. Total scores of 0-6 indicate 'none to mild depression' and scores of 16-24 indicate 'severe depression'. Data from participant visits at baseline, 3 months, 9 months, 15 months and 21 months were combined and averaged to calculate a single value.
Time Frame: Up to 21 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 10 | 9
score on a scale | 4.75 (4.98) | 5.7 (4.62) | 4.38 (5.12)

7. Secondary Outcome: The Severity of Anxiety as Measured by the Adapted New Zealand Health Promotion Agency Anxiety Self-Test
Description: The adapted New Zealand Health Promotion Agency Anxiety Self-Test is an 8 question self-administered questionnaire that scores patient-reported symptoms of anxiety. The possible score for each question ranges from 0-3. The total questionnaire score range is 0-24. Total scores of 0-8 indicate 'none to mild anxiety' and scores of 16-24 indicate 'severe anxiety'. Data from participant visits at baseline, 3 months, 9 months, 15 months and 21 months were combined and averaged to calculate a single value.
Time Frame: Baseline to 21 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 7 | 10 | 9
score on a scale | 5.0 (6.88) | 3.55 (3.32) | 5.61 (7.25)

8. Secondary Outcome: The Percentage of Change in Forced Vital Capacity (FVC) Measured by Spirometry
Description: The percentage of change in home-measured forced vital capacity (FVC) compared to clinic-measured FVC via spirometry
Time Frame: Baseline to 21 months
Population: Incomplete data was collected due to non-standardized practices (e.g., no standard processes in place for how data was collected, formatted, or reported). Data not collected includes: Usual Care: Missing data from 7 participants / Telenursing: Missing data from 10 participants / Telenursing and Remote Monitoring: Missing data from 9 participants. Exhaustive efforts were made to obtain the missing data, but the original PI has left and it is nonexistent in the EDC and cannot be located elsewhere.
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 21 months
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) | Telenursing | Telenursing and Remote Monitoring
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care of Idiopathic Pulmonary Fibrosis (IPF) (N=7) | Telenursing (N=10) | Telenursing and Remote Monitoring (N=9)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to the original PI leaving the institution. The new PI never enrolled any participants and the study was closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03562247/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT03562247/ICF_001.pdf